CLINICAL TRIAL: NCT01601301
Title: A Post-Market Prospective Evaluation of the Performance and Safety of the Ellipse PRECICE Intramedullary Limb Lengthening System
Brief Title: Post-Market Study of the Ellipse PRECICE Intramedullary Limb Lengthening System
Acronym: PINS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ellipse Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR0035
Record Dates: First submitted 2012-05-14; First posted 2012-05-18 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Limb Length Discrepancy
Keywords: Limb; Lengthening; PRECICE; Ellipse; Technologies; Distraction; Osteogenesis; Femur; Tibia; Intramedullary; Nail; Device; Medical; Orthopedic; Implant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PRECICE System (Experimental)
  Interventions: Device: PRECICE System

INTERVENTIONS:
Device: PRECICE System — Lenthening of either the tibia or femur with the PRECICE System.

SUMMARY:
The purpose of this study is to obtain post market performance and safety data of the Ellipse PRECICE Intramedullary Limb Lengthening System for subjects undergoing unilateral limb lengthening.

DETAILED DESCRIPTION:
Subject data will be reviewed at the following visits:

* Preoperative
* Operative
* Every 7 to 14 days through Distraction Phase
* Every 4 to 6 weeks through Consolidation Phase
* 6-Month Post-Consolidation
* 12-Month Post-Consolidation
* 18-Month Post-Consolidation
* 24-Month Post-Consolidation

ELIGIBILITY:
Inclusion Criteria:

* Leg length discrepancy ≥ 1.5 cm and ≤ 6.5 cm due to short femur or tibia
* Weight ≤ 114 kg if implanted with the 10.7 mm or 12.5 mm diameter nail, or ≤ 57 kg if implanted with the 8.5 mm diameter nail
* Skeletally mature
* Intramedullary canal without offset
* Tibia or femur sufficient to contain the implant
* Availability, willingness, and sufficient cognitive awareness to comply with protocol procedures and schedule
* Must sign informed consent to permit the use of personal health data

Exclusion Criteria:

* Active infection or previous history of deep infection in the involved bone
* Metal allergies or sensitivities to the components of the device
* Distance from the nearest convenient external surface of the treated limb to the intramedullary canal > 38 mm for the 8.5 mm PRECICE nail, > 51 mm for the 10.7 mm PRECICE nail, or > 76 mm for the 12.5 mm PRECICE nail
* Significant range of motion deficit of the adjacent joints
* Patients with a pacemaker, implanted cardiac defibrillator, or any other electronic or magnetic implant
* Patients who require an MRI during implantation
* Non-union
* Impassable or obstructed intramedullary canal
* Significant angular deformity that prevents device placement
* Cannot bear weight on the contralateral limb
* Procedural osteotomy cannot be made in an appropriate location
* Deformities that require multilevel osteotomies or bi-lateral implantation at the time of study index surgery
* Systemic bone disease
* Pregnant or nursing women
* Inadequate vascularity or evidence of vascular disease or peripheral neuropathy
* Malignancies or tumors in the involved bone
* Patient is a drug abuser
* Open wounds or ulcers that could compromise treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-07; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Distraction Control: actual distraction rate vs. target distraction rate | Postoperatively, every 7-10 days up until the subject's distraction regimen is complete, an expected average of 33 days

SECONDARY OUTCOMES:
Bone Union | Following completion of the subject's distraction regimen, every 4-6 weeks until the subject's treated limb is evaluated as consolidated, an expected average of 66 days
Pain | Up to 24 months post-consolidation of the treated limb, an expected total average of 29 months
  Pain measured by the SF-36v2, American Academy of Orthopaedic Surgeons Lower Limb Outcomes Questionnaire, and medication use.
Healing Index | Up to 24 months post-consolidation of the treated limb, an expected total average of 29 months
  The total treatment period with the PRECICE System in situ, divided by the length of bone growth in centimeters.
Number of days to complete lengthening | Postoperatively, every 7-10 days up until the subject's distraction regimen is complete, an expected average of 33 days
Number of days to complete full weight bearing | Up to an expected average of 99 days.
Number of days to full consolidation | Following completion of the subject's distraction regimen, every 4-6 weeks until the subject's treated limb is evaluated as consolidated, an expected average of 66 days
Adverse Events | Up to 24 months post-consolidation of the treated limb, an expected total average of 29 months
Device-related complications | Up to 24 months post-consolidation of the treated limb, an expected total average of 29 months
Procedure-related complications | Up to 24 months post-consolidation of the treated limb, an expected total average of 29 months

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A Green, MD, Principal Investigator — University of California, Irvine
Locations (6):
- United States (6):
  - Loma Linda University, Loma Linda, California
  - Nemours Children's Hospital, Orlando, Florida
  - Paley Advanced Limb Lengthening Institute, West Palm Beach, Florida
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Hospital for Special Surgery, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio